CLINICAL TRIAL: NCT06677333
Title: The Effect of Increasing Dietary Protein on the Gut Microbiota
Brief Title: The Effect of Increasing Dietary Protein on the Gut Microbiome and Its Metabolites
Acronym: PSGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5008
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-09

CONDITIONS: Health Adults
Keywords: gut microbiota; dietary protein; gut metabolites; gut metabolome; dietary purines; gut microbiome
MeSH Terms: interventions — Whey Proteins; Pea Proteins

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to consume 50 g of whey or pea protein for seven days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whey protein supplement (Experimental): This group of participants will consume 50 g of whey protein supplement daily.
  Interventions: Other: Whey Protein
- Pea protein supplement (Experimental): This group of participants will consume 50 g of pea protein supplement daily.
  Interventions: Other: Pea protein

INTERVENTIONS:
Other: Whey Protein — This intervention will add 50 g of a whey or pea protein supplement to their usual dietary intake.
  Arms: Whey protein supplement
Other: Pea protein — This intervention will add 50 g of a pea protein supplement to their usual dietary intake.
  Arms: Pea protein supplement

SUMMARY:
This study will determine the effect of dietary protein not absorbed in the small intestine on the bacteria in the large intestine and the metabolites those bacteria produce when they break down the protein. The three specific goals are:

1. Determine if increasing dietary protein increases the purine breakdown product, allantoin, as observed in our previous study.
2. Establish a model to examine the effect of dietary protein on the gut microbiota and metabolites.
3. Identify gut bacteria and metabolite changes that occur with increased consumption of animal (whey) or plant (pea) protein sources.

DETAILED DESCRIPTION:
Healthy male and female participants were recruited following specific inclusion/exclusion criteria. Participants were excluded if they 1) were less than 25 years of age, 2) consumed pre or probiotics in the last week, 3) had taken any antibiotics in the last three months, 4) were taking any prescribed medicines for a chronic disease such as diabetes, hypertension, cancer, anxiety, depression, or GI-related diseases. and 4) had taken any laxatives or antidiarrhea inhibitors in the last week. The study design was pre/post, with each person serving as their own control. Interested participants were randomly assigned to one of two study groups: 50 g whey protein supplement or 50 g pea protein supplement. They were asked to consume the supplement along with their usual dietary intake. Participants were located within the contiguous USA and were sent a fecal collection kit, the protein supplement, and a shaker bottle using overnight shipping. We used the fecal collection kit developed by the Biocollective. A fecal sample was collected before and after the participant consumed the protein supplement daily for seven days. At both time points, the participants were asked to recall the foods they ate during the previous 24 hours using ASA24-2020, provide information on their physical activity (International Physical Activity Questionnaire, IPAQ), and answer questions about the stool sample they collected. The stool sample will be analyzed for the microbes and metabolites present. These will be correlated with the dietary protein they consume.

ELIGIBILITY:
Inclusion Criteria:

* 25 years old or older
* male or female
* located in the contiguous United States

Exclusion Criteria:

* Taken any prebiotics in the last week
* Taken any probiotics in the last week
* Taken any prescription medications other than oral contraceptives
* Taken antibiotics sometime in the last three months
* Taken any diarrhea inhibitors in the last week
* Taken any laxatives in the last week
* Taken any dietary supplement(s)
* Diagnosed with cancer
* Diagnosed with an inflammatory disease of the GI tract, such as irritable bowel disease
* Experienced long-haul COVID fatigue
* Were physically inactive (<600 METS per week)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Fecal allantoin | A fecal sample is collected before and after consuming a protein supplement (pea or whey) for seven days.
  A cross-sectional study the investigators conducted found that healthy individuals who reported consuming, on average, 150 gms of protein daily had a higher fecal allantoin. This study is a pre/post-randomized controlled trial to confirm that observation. It will determine if consuming 50 gms more protein daily increases fecal allantoin.

SECONDARY OUTCOMES:
Changes in fecal bacterial species before and after increasing dietary protein intake (pea or whey) by 50 grams for seven days | A fecal sample is collected before and after consuming a protein supplement (pea or whey) for seven days.
  The relative abundance of fecal bacterial species before and after consuming an additional 50 grams of pea or whey protein above the participant's usual dietary protein intake for seven days will be compared for each group to identify which species have significantly increased or decreased.
Changes in fecal metabolites before and after increasing dietary protein intake (pea or whey) by 50 grams for seven days | A fecal sample is collected before and after consuming a protein supplement (pea or whey) for seven days.
  The intensity of fecal metabolites will be measured using mass spectrometry. The difference before and after consuming an additional 50 grams of pea or whey protein above the participant's usual dietary protein intake for seven days will be compared for each group to identify those metabolites that have significantly increased or decreased.

CONTACTS AND LOCATIONS:
Overall Officials: Lauri O. Byerley, PhD, Principal Investigator — APUS/LSUHSC
Locations (1):
- Louisiana State University Health Sciences Center New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be submitted six months after article publication. Qualified researchers engaged in independent scientific research can request access to this study's IPD, which will be provided following the review and approval of a research proposal, Statistical Analysis Plan (SAP), and execution of a Data Sharing Agreement (DSA). Data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis. For more information or to submit a request, please contact lbyerl@lsuhsc.edu.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted six months after article publication and will be accessible for up to 24 months.
Access Criteria: Qualified researchers engaged in independent scientific research can request access to this study's IPD, which will be provided following the review and approval of a research proposal, Statistical Analysis Plan (SAP), and execution of a Data Sharing Agreement (DSA). D